CLINICAL TRIAL: NCT04289376
Title: Quiet Eye Duration in Baseball
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Nicklaus Fogt, Professor, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2019H0403
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Gaze Tracking
Keywords: Sports

STUDY DESIGN:
Intervention Model Description: There is no intervention or treatment in this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gaze tracking (Other): No intervention. Monitor gaze as subjects watch a video
  Interventions: Other: Gaze tracking - no intervention

INTERVENTIONS:
Other: Gaze tracking - no intervention — Monitor gaze as subjects watch a video

SUMMARY:
The purpose of this study is to measure the gaze movements of individuals as they watch videos of a baseball pitcher throwing pitches. The goal will be to determine whether there is an anticipatory movement to the location where the ball is released, and whether this anticipatory movement occurs in experienced baseball players more commonly than in inexperienced players.

DETAILED DESCRIPTION:
20 subjects between 18 and 40 years of age (males and females) will participate. 10 subjects will be required to have experience in baseball or softball at the high school level or above within the last 10 years. A further 10 subjects will be recruited who did not have baseball experience at or above the high school level. Upon entering the laboratory, the experiment will be explained to the subjects. Subjects will be consented. Then, the subject's visual acuity and stereoacuity (depth perception) will be measured.

If subjects continue on to the experiment, they will also be asked to complete a short survey on previous baseball experience.

Subjects will stand in a batting stance facing a projector screen. They will then participate in trials in which they mimic batting a ball thrown by a pitcher. Six different pitch videos will be shown. The subjects will act as if they are batting the ball (no bat swing will occur) for each video. The movement of the subject's eye will be tracked using an eye tracker.

ELIGIBILITY:
Inclusion Criteria:

* 20/20 visual acuity in each eye Stereoacuity of 40 arc seconds are better

Exclusion Criteria:

* 20/25 or worse visual acuity in either eye Stereoacuity less than 40 arc seconds

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Quiet eye duration | 60 minutes
  Duration over which the gaze remains stable

CONTACTS AND LOCATIONS:
Overall Officials: Nick F Fogt, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No